CLINICAL TRIAL: NCT05676619
Title: Reliability of 3D Foot Scanner for Use in Diabetes Fit Evaluation and Footwear Design
Brief Title: 3D Foot Scanner Reliability for Footwear Fit and Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0865
Record Dates: First submitted 2022-12-19; First posted 2023-01-09 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Complications
Keywords: 3D foot scan; 3D foot scanner; foot scan; reliability; repeatability
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single cohort of healthy volunteers (Other): Single cohort of healthy volunteers
  Interventions: Device: 3D foot scanner

INTERVENTIONS:
Device: 3D foot scanner — Reliability of 3D foot scanner during repeated scans

SUMMARY:
The investigators will carry out a proof-of-concept study in 20 adult healthy male and female volunteers in order to: assess a 3D foot scanner's reliability. Specifically, the investigators will assess its variability during repeated foot scans of the same subject's foot. Three repeated foot scans will be carried out by two different examiners to measure intrarater and interrater reliability (Intraclass Correlation Coefficient

DETAILED DESCRIPTION:
Evidence of reliability is essential for use of a 3D foot scanner in diabetes footwear fit evaluation and orthopaedic footwear design. The investigators will carry out a proof-of-concept study in 20 healthy adult male and female volunteers in order to: assess the 3D foot scanner's reliability. Specifically, the investigators will assess its variability during three repeated foot scans of the same subject's foot. Three half weightbearing foot scans will be carried out by two different examiners to measure intrarater and interrater reliability (Intraclass Correlation Coefficient).

The investigators will carry out a proof-of-concept study in 20 healthy adult male and female volunteers (10 each) in order to assess the Elinvision 3D foot scanner's (i) intra-rater reliability through repeated foot scans (3 times each) and (ii) inter-rater reliability of these scans as carried out by two independent examiners whilst participants are half weightbearing to establish adequate reliability (0.80+ ICC) for use in subsequent diabetes footwear fit assessment and orthopaedic footwear design and manufacture.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18 years or over
* Able to walk unaided
* Able to walk up steps (the 3D scanner requires a small step on to the device to enter the correct position for measurement)
* Willingness and capacity to participate in the study and to sign the informed consent form

Exclusion Criteria:

* Diabetes mellitus diagnosis
* Inability to ambulate independently without walking aids
* No obvious foot deformities
* No history of foot surgery
* No pain, injuries or medical conditions affecting the legs or lower back
* Any issues around balance (participants must remain standing in position for the approximately fifteen seconds required to obtain the 3D scan of their feet)
* Health conditions that impact foot morphology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
Intrarater reliability (Intraclass Correlation Coefficient) of 3D foot scans repeated at baseline (change) | Repeated scans at baseline
  (i) Intrarater reliability (Intraclass Correlation Coefficient) based on three scans of the same subject's foot whilst half-weightbearing carried out by the same 'rater' i.e. person using the 3D foot scanner;
Interrater reliability (Intraclass Correlation Coefficient) of 3D foot scans repeated at baseline (change) | Repeated scans at baseline
  (ii) Interrater reliability (Intraclass Correlation Coefficient) based on three scans of the same subject's foot first by one rater (as above) and then by a second rater

CONTACTS AND LOCATIONS:
Overall Officials: Petra J Jones, Principal Investigator — University Hospitals, Leicester
Locations (1):
- Leicester General Hospital, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers